CLINICAL TRIAL: NCT03668522
Title: Clinical Research of the Molecular Phenotype Distribution of H3F3AK27M in Spinal Glioma and Its Impact on TMZ Chemoradiotherapy
Brief Title: Clinical Research of H3F3AK27M in Spinal Glioma and Its Impact on TMZ Chemoradiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Yuntao Lu, adjunct professor, Southern Medical University, China
Other Study IDs: SouthernMUC Neurospine-1
Record Dates: First submitted 2018-09-03; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Spinal Tumor
Keywords: H3F3AK27M
MeSH Terms: conditions — Spinal Cord Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children: age<=17
  Interventions: Other: Genetic testing
- adult: age>17
  Interventions: Other: Genetic testing

INTERVENTIONS:
Other: Genetic testing — To determine whether H3F3AK27M exist in spinal glioma

SUMMARY:
H3F3AK27M may be a feature of primary spinal cord glioma and affect the outcome and prognosis of TMZ chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Surgical treatment and pathological confirmation of spinal glioma in our department and is the first case without any treatment before operation.

Exclusion Criteria:

* The tumor is recurrent or has been treated before operation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgical treatment and pathological confirmation of spinal glioma in our department.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
positive | through study completion, an average of 1 year
  positive of H3F3AK27M

CONTACTS AND LOCATIONS:
Overall Officials: Lu Yuntao, M.D., Ph.D, Study Chair — Nanfang Hospital Neurosurgery Department
Locations (1):
- Nan fang hospital, Southern medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided